CLINICAL TRIAL: NCT03429855
Title: Effectiveness of Bobath Based Trunk Training on in Acute Stroke Patients: a Randomized Controlled Trial
Brief Title: Bobath Approach for Trunk Control in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ayla fil balkan, assoc prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-16073
Record Dates: First submitted 2018-01-22; First posted 2018-02-12 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute
Keywords: Physiotherapy; Trunk control; Bobath concept; Stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Bobath based trunk exercises
  Interventions: Other: trunk training
- control group (Other): conventional physiotherapy approaches
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: trunk training — Bobath based trunk training
  Arms: study group
Other: physiotherapy — conventional physiotherapy
  Arms: control group

SUMMARY:
In stroke patients, the impairment of the trunk affects many functions negatively. For this reason training of the trunk is necessary in the early period. Taking into account of literature, various approaches have been used to improve sitting balance and trunk control such as conventional physiotherapy for stroke patients . Bobath concept is another method used for stroke rehabilitation. When the studies about stroke rehabilitation are investigated, it is seen that most of the studies included only chronic patients and Bobath concept did not adequately take place in literature about trunk training. The aim of this study is to determinate effectiveness of the Bobath based trunk training on trunk control in acute stroke patients.

DETAILED DESCRIPTION:
In stroke patients, the impairment of the trunk affects many functions negatively. For this reason training of the trunk is necessary in the early period. Taking into account of literature, various approaches have been used to improve sitting balance and trunk control such as conventional physiotherapy for stroke patients . Bobath concept is another method used for stroke rehabilitation. Trunk control is an important issue in the Bobath approach since the acute period. It seems that the Bobath method, which includes both approaches to increase postural control and sitting, as well as applications to increase the sensation, seems to be an appropriate method to improve body control in stroke patients. When the studies about stroke rehabilitation are investigated, it is seen that most of the studies included only chronic patients and Bobath concept did not adequately take place in literature about trunk training in acute stroke. The aim of this study is to determinate effectiveness of the Bobath based trunk training on trunk control in acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* patients scoring ≥14 on Glasgow Coma Scale and Mini Mental Test>24

Exclusion Criteria:

* patients scoring <14 on Glasgow Coma Scale
* patients with recurrent strokes
* patients with orthopedic or neurological disorders (other than strokes) that might affect their motor performance

Ages: 42 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale (by Verheyden) | Change from Baseline the scale score at 20th days in hospital
  It consists of 3 subscales of static and dynamic sitting balance and trunk coordination, scored up to 7, 10, and 6 points, respectively.The total scores range between 0 and 23 points, where a higher score indicates better truncal function.
Trunk Control Test | Change from Baseline the scale score at 20th days in hospital
  The test consists of four items which are assessed on a 3-point ordinal scale.The total score for the Trunk Control Test ranges from minimum 0 to maximum 100 points, a higher score indicating a better performance.
Motor Assessment Scale | Change from Baseline the scale score at 20th days in hospital
  It contains three items assessing trunk performance. Each item is scored on a 7-point ordinal scale, a higher score indicating a better performance.
Berg Balance Scale | Change from Baseline the scale score at 20th days in hospital
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. It is a valid instrument used for evaluation of the effectiveness of interventions and for quantitative descriptions of function in clinical practice and research. The BBS has been evaluated in several reliability studies.
independently sitting time | Change from Baseline sitting time at 20th days in hospital
  Sitting with back unsupported without using hands but feet supported on floor.

SECONDARY OUTCOMES:
Glasgow Coma Scale | Baseline, on 7th, 10th and 20th days during the treatment
  It assessed the initial and subsequent level of consciousness in a person after a brain injury. Mild head injuries are generally defined as those associated with a Glasgow Coma scale score of 13-15.
Modified Rankin Scale | Baseline, on 7th, 10th and 20th days during the treatment
  The Modified Rankin Scale (MRS) is the most commonly used to evaluate the degree of disability or dependence in the daily activities of people who have suffered a stroke. It describes "global disability" with a focus on mobility. The MRS is an ordered scale coded from 0 (no symptoms at all) through 5 (severe disability) 6 (death).
The Functional Independence Measure (FIM) | Baseline, on 7th, 10th and 20th days during the treatment
  The Functional Independence Measure (FIM) evaluates self-care, sphincter control, mobility, locomotion, communication, and social cognition. The FIM item scores range from 1 (total assistance required) to 7 (complete independence). A higher score indicates a greater degree of independence with regard to daily living activities. This subscale has good psychometric properties for stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Fil Balkan, Asst. Prof, Principal Investigator — Hacettepe University; Ali Naim Ceren, MSc, Study Chair — Hacettepe University; Ceren Saban, MSc, Study Chair — Eskişehir Osmangazi University Health Application and Research Hospital; Yeliz Salcı, Asst. Prof, Study Chair — Hacettepe University; Hilal Keklicek, Asst. Prof, Study Chair — Trakya University; Kadriye Armutlu, Prof Dr, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] Verheyden G, Nieuwboer A, Van de Winckel A, De Weerdt W. Clinical tools to measure trunk performance after stroke: a systematic review of the literature. Clin Rehabil. 2007 May;21(5):387-94. doi: 10.1177/0269215507074055. PMID 17613559
- [Background] Collin C, Wade D. Assessing motor impairment after stroke: a pilot reliability study. J Neurol Neurosurg Psychiatry. 1990 Jul;53(7):576-9. doi: 10.1136/jnnp.53.7.576. PMID 2391521
- [Background] Carr JH, Shepherd RB, Nordholm L, Lynne D. Investigation of a new motor assessment scale for stroke patients. Phys Ther. 1985 Feb;65(2):175-80. doi: 10.1093/ptj/65.2.175. PMID 3969398
- [Background] Bank J, Charles K, Morgan P. What is the effect of additional physiotherapy on sitting balance following stroke compared to standard physiotherapy treatment: a systematic review. Top Stroke Rehabil. 2016 Feb;23(1):15-25. doi: 10.1179/1945511915Y.0000000005. Epub 2015 Jun 18. PMID 26086177
- [Background] Kilinc M, Avcu F, Onursal O, Ayvat E, Savcun Demirci C, Aksu Yildirim S. The effects of Bobath-based trunk exercises on trunk control, functional capacity, balance, and gait: a pilot randomized controlled trial. Top Stroke Rehabil. 2016 Feb;23(1):50-8. doi: 10.1179/1945511915Y.0000000011. Epub 2015 Aug 10. PMID 26260878
- [Background] Benito Garcia M, Atin Arratibel MA, Terradillos Azpiroz ME. The Bobath Concept in Walking Activity in Chronic Stroke Measured Through the International Classification of Functioning, Disability and Health. Physiother Res Int. 2015 Dec;20(4):242-50. doi: 10.1002/pri.1614. Epub 2014 Dec 4. PMID 25475602
- [Background] Cabanas-Valdes R, Cuchi GU, Bagur-Calafat C. Trunk training exercises approaches for improving trunk performance and functional sitting balance in patients with stroke: a systematic review. NeuroRehabilitation. 2013;33(4):575-92. doi: 10.3233/NRE-130996. PMID 24018373